CLINICAL TRIAL: NCT03996915
Title: Evaluation of Halitosis in Adult Patients After Treatment With Photodynamic Therapy Associated With Periodontal Treatment: Protocol for a Randomized, Controlled Single Blinded Trial With 3-month Follow up
Brief Title: Evaluation of Halitosis After Treatment With Photodynamic Therapy Associated With Periodontal Treatment
Acronym: Halitosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Phd, clinical professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Halitosis healthy patients
Record Dates: First submitted 2019-06-22; First posted 2019-06-25 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2019-12

CONDITIONS: Halitosis
Keywords: photodynamic therapy; periodontal disease; randomized controlled clinical study
MeSH Terms: conditions — Halitosis; Periodontal Diseases | interventions — Ultraviolet Therapy

STUDY DESIGN:
Intervention Model Description: Bio-equivalence Study Enrollment:40
Who Masked: Investigator
Masking Description: single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental PDT group (Experimental): G1-20 patients Photodynamic therapy with methylene blue as photosensitizer device irradiation with low intensity laser (wave length = 660 nm) 9 J (Joules) per point (6 points) and radiant 90 seconds. Photosensitiser (PS) will be applied in sufficient quantity to cover the middle third and back of the tongue and wait for 5 minutes.Six points with the distances of 1 cm between them will be irradiated.
  Interventions: Device: Pdt Photodynamic Therapy
- control tongue scrapper group (Active Comparator): G2-20 patients Tongue scrapping will be performed by the same operator in all patients. Posterior -anterior movements will be performed with the scrapper over the lingual dorsum in order to promote the mechanical removal of tongue coating
  Interventions: Other: tongue scrapper

INTERVENTIONS:
Device: Pdt Photodynamic Therapy — device irradiation with low intensity laser (wave length = 660 nm) 9 J (Joules) per point(6 points) and radiant 90 seconds PS will be applied in sufficient quantity to cover the middle third and back of the tongue and wait for 5 minutes.six points with the distances of 1 cm between them will be irradiated.
  Arms: experimental PDT group
Other: tongue scrapper — Tongue scrapping will be performed by the same operator in all patients. Posterior -anterior movements will be performed with the scrapper over the lingual dorsum. in order to promote the mechanical removal of tongue coating
  Arms: control tongue scrapper group

SUMMARY:
The aim of this randomized, controlled clinical trial was to treat oral halitosis in healthy adults with photodynamic therapy associated with periodontal treatment and follow them up for 3 months. The participants with halitosis will be randomized into two groups: G1-treatment with photodynamic therapy or G2-cleaning of the tongue with a tongue scraper . Halitosis were evaluated measuring volatile sulfur compounds using gas chromatography After the treatments, a second evaluation will be performed, along with a microbiological analysis (qPCR) for the identification of the bacteria T. denticola

DETAILED DESCRIPTION:
Halitosis is an unpleasant odor that emanating from the mouth. A recent metanalysis shows worldwide trend towards a rise in halitosis prevalence. Studies show halitosis returns in a week after treatment with photodynamic therapy (PDT). Probably, bacteria residing in the periodontal sulcus could recolonize the dorsum of the tongue. To date, there are no study in adult population that associate halitosis and periodontal treatment with follow-up evaluation. The aim of this randomized, controlled clinical trial was to treat oral halitosis in healthy adults with photodynamic therapy associated with periodontal treatment and follow them up for 3 months. The participants (n=40) with halitosis will be randomized into two groups: G1-treatment with photodynamic therapy (n = 20) or G2-cleaning of the tongue with a tongue scraper (n = 20). Halitosis were evaluated measuring volatile sulfur compounds using gas chromatography After the treatments, a second evaluation will be performed, along with a microbiological analysis (qPCR) for the identification of the bacteria T. denticola. The evaluation of halitosis and the microbiological analysis will be repeated. After that, patients will receive periodontal treatment. The participants will return after 1 week and three months for an additional evaluation. Quality of life will be measured by Oral Health Impact Profile (OHIP-14) Comparisons will be made with ANOVA test, with the level of significance of 5 %. This protocol will determine the effectiveness of phototherapy regarding the reduction of halitosis in adults.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* with at least 10 teeth
* Periodontal screening and recording (PSR) 0, 1 or 2
* without any changes in the anatomy of the back of the tongue (geographical or fissured tongue)
* positive halitosis (SH2 level higher than 112 ppb).

Exclusion Criteria:

* smokers
* ex-smokers for less than 5 years
* patients with hypersensitivity to the photosensitizer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
halitosis measurement (gas chromatography test) | through study completion on average of one year
  The portable Oral Chroma will be used for the assessment of halitosis. Oral air collection will follow the manufactured guide lines (Oral Chroma Manual Instruction). A syringe will be placed in the patient's mouth with the plunger completely inserted and the participant will breathe through the nose with the mouth closed for one minute.The plunger will then be withdrawn to fill the chamber with air. This procedure will be repeated. The gas injection needle will be placed on the syringe and the plunger will be adjusted to 0.5 ml. This air will be injected into the input of the device in a single motion. This procedure will be done before, immediately after PDT or scraper and after periodontal treatment.

SECONDARY OUTCOMES:
microbiological analysis | through study completion on average of one year
  collecting biofilm sample from the region of the lingual dorsum with swab and identification of the bacteria P. gingivalis and T. denticola. Sample will be transferred to sterile tubes with ethylenediaminetetraacetic acid (tris-EDTA). The analysis will be performed by PCR (polymerase Chain reaction) real time

CONTACTS AND LOCATIONS:
Overall Officials: Anna Carolina rt Horliana, phd, Principal Investigator — Nove de Julho University
Locations (1):
- Nove de Julho University (UNINOVE), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] da Silva T, da Silva FC, Gomes AO, Viana AO, Goncalves MLL, Rodrigues MFSD, Horliana ACRT, da Silva DFT, Chavantes MC, Fragoso YD, Branco LP, Motta LJ, Fernandes KPS, Mesquita-Ferrari RA, Bussadori SK. Effect of photobiomodulation treatment in the sublingual, radial artery region, and along the spinal column in individuals with multiple sclerosis: Protocol for a randomized, controlled, double-blind, clinical trial. Medicine (Baltimore). 2018 May;97(19):e0627. doi: 10.1097/MD.0000000000010627. PMID 29742699
- [Background] Sobral APT, Godoy CLH, Fernandes KPS, Bussadori SK, Ferrari RAM, Horliana ACRT, Monken SF, Motta LJ. Photomodulation in the treatment of chronic pain in patients with temporomandibular disorder: protocol for cost-effectiveness analysis. BMJ Open. 2018 May 5;8(5):e018326. doi: 10.1136/bmjopen-2017-018326. PMID 29730613
- [Background] da Cunha Moraes G, Vitoretti LB, de Brito AA, Alves CE, de Oliveira NCR, Dos Santos Dias A, Matos YST, Oliveira-Junior MC, Oliveira LVF, da Palma RK, Candeo LC, Lino-Dos-Santos-Franco A, Horliana ACRT, Gimenes Junior JA, Aimbire F, Vieira RP, Ligeiro-de-Oliveira AP. Low-Level Laser Therapy Reduces Lung Inflammation in an Experimental Model of Chronic Obstructive Pulmonary Disease Involving P2X7 Receptor. Oxid Med Cell Longev. 2018 Mar 4;2018:6798238. doi: 10.1155/2018/6798238. eCollection 2018. PMID 29686745
- [Derived] Romero SDS, Schalch TO, do Vale KL, Ando ES, Mayer MPA, Feniar JPG, Fernandes KPS, Bussadori SK, Motta LJ, Negreiros RM, Tempestini Horliana ACR. Evaluation of halitosis in adult patients after treatment with photodynamic therapy associated with periodontal treatment: Protocol for a randomized, controlled, single-blinded trial with 3-month follow up. Medicine (Baltimore). 2019 Sep;98(39):e16976. doi: 10.1097/MD.0000000000016976. PMID 31574796